CLINICAL TRIAL: NCT07389356
Title: Rituximab, Ifosfamide, Mitoxantrone Liposome, Etoposide (Modified R-MINE) Regimen vs. Rituximab, Gemcitabine and Oxaliplatin (R-GemOx) Regimen in the Treatment of Late Relapsed Diffuse Large B-cell Lymphoma: A Multicenter, Open, Randomized, Controlled, Phase II Study
Brief Title: Modified R-MINE Regimen vs. R-GemOx Regimens on the Treatment of Late Relapsed DLBCL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DED-DLBCL-K16
Record Dates: First submitted 2025-12-17; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: DLBCL - Diffuse Large B Cell Lymphoma
Keywords: DLBCL; Mitoxantrone Hydrochloride liposomal
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- modified R-MINE (Experimental)
  Interventions: Drug: Rituximab+Ifosfamide+Mesna+Mitoxantrone hydrochloride liposome+Etoposide
- R-GemOx (Active Comparator)
  Interventions: Drug: Rituximab+Gemcitabine+Oxaliplatin

INTERVENTIONS:
Drug: Rituximab+Ifosfamide+Mesna+Mitoxantrone hydrochloride liposome+Etoposide — Rituximab 375 mg/m^2, d0; Ifosfamide 1.33 g/m^2, d1-3 (equal dose of mesna rescue); Mitoxantrone hydrochloride liposome 12mg/m^2, d1; Etoposide 65 mg/m^2, d1-3; Every 21 days as one cycle, and 4 cycles were planned.
  Arms: modified R-MINE
Drug: Rituximab+Gemcitabine+Oxaliplatin — Rituximab 375 mg/m^2, d0; Gemcitabine 1000 mg/m^2, d1; Oxaliplatin 100 mg/m^2, d1; Every 21 days as one cycle, and 4 cycles were planned.
  Arms: R-GemOx

SUMMARY:
This study was a multicenter, open, randomized controlled, phase II clinical study. Is expected in 70 cases of late relapsed diffuse large B cell lymphoma, were randomly assigned to receive mitoxantrone liposomes modified R - MINE plan or R - GemOx treatment. Each cycle was 3 weeks (21 days) for a total of 4 cycles. Subjects assigned to each signed informed consent to screening, screening, in the center of the study determined in accordance with the order signed informed consent. Before the start of the trial, the number of random seeds was set by the statistician, and the block randomization method was used to generate the subject random table using R 4.3.3 (or above). The random ratio between the modified R-mine group and the R-Gemox group was 1:1. After the investigator determined that the subjects were screened successfully, the subjects were randomly numbered according to the order in which the eligible subjects were screened successfully. The intervention was performed by the principal investigator or by someone designated by the principal investigator. Study includes screening period (the first 28 days), treatment period (plan 4 cycles, treatment after 2 cycles enhanced CT/MRI or PET - CT mid-term efficacy, PET - CT curative effect evaluation) after treatment, follow-up (follow-up curative effect, safety and survival follow-up follow-up). Participants provided written informed consent and underwent baseline examinations during the screening period. Participants who met the inclusion criteria and none of the exclusion criteria entered the treatment period. All the study participants completed protocol-specified examinations during the course of treatment to observe efficacy and safety. The end of the treatment period was followed by the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* They voluntarily participated in the study and signed the informed consent.
* Age 18 or higher;
* Expected survival time for 3 months or more;
* The histopathological diagnosed late relapsed (> 12 months) diffuse large B cell lymphoma;
* Must have at least a Lugano 2014 standard can be evaluation or measurable lesions: lymph node lesions, measurable lymph nodes should be diameter > 1.5 cm; Non-lymph node lesions, measurable extranodal lesions should be diameter > 1.0 cm;
* ECOG score 0 to 2 points;
* Bone marrow function: neutrophil count >= 1.5 x 10^9 / L, platelet count >= 75 x 10^9 / L, and hemoglobin >= 80 g/L (neutrophil count may be extended to >= 1.0 x 10^9 / L, the platelet count can be extended to >= 50 x 10^9 / L, and hemoglobin can be extended to >= 75 g/L in patients with bone marrow involvement);
* Liver and kidney function: serum creatinine acuities were <= 1.5 times the upper limit of normal (ULN) value; AST and ALT <= 2.5 times the ULN(<= 5 times the upper limit of normal in patients with liver invasion); Total bilirubin <= 1.5 times the ULN (<= 3 times the upper limit of normal in patients with liver invasion);
* Blood coagulation function: International standardization Ratio (International Normalized thewire, INR) <= 1.5 x ULN; Prothrombin Time (PT), Activated PartialThromboplastin Time (APTT) <= 1.5×ULN (unless receiving anticoagulant therapy, And PT and APTT at screening were within the expected range for anticoagulant therapy).

Exclusion Criteria:

* Previous history of antitumor therapy meeting any of the following conditions:

  1. Prior treatment with mitoxantrone or liposomal mitoxantrone;
  2. Prior treatment with doxorubicin or other anthracyclines, with a total cumulative doxorubicin dose >360 mg/m² (for other anthracyclines, 1 mg of doxorubicin is equivalent to 2 mg of epirubicin);
  3. Prior autologous hematopoietic stem cell transplantation within 100 days before the first dose, or a history of allogeneic hematopoietic stem cell transplantation;
  4. Prior antitumor therapy (including chemotherapy, targeted therapy, hormone therapy, traditional Chinese medicine with antitumor activity, etc.) or participation in other clinical trials involving investigational drugs within 4 weeks or 5 half-lives (whichever is shorter) before the first dose of the study drug.
* Hypersensitivity to any study drug or its components;
* Uncontrolled systemic diseases (e.g., progressive infections, uncontrolled hypertension, diabetes, etc.);
* Cardiac function and diseases meeting any of the following conditions:

  1. Long QTc syndrome or QTc interval >480 ms;
  2. Complete left bundle branch block, complete right bundle branch block with left anterior fascicular block, type II second-degree or third-degree atrioventricular block;
  3. Severe, uncontrolled arrhythmia requiring medication;
  4. New York Heart Association Class ≥ III;
  5. History of acute myocardial infarction, unstable angina, severe unstable ventricular arrhythmia, or any other arrhythmia requiring treatment within 6 months before enrollment; history of clinically significant pericardial disease; or electrocardiographic evidence of acute ischemic or active conduction system abnormalities.
* Active hepatitis B or C infection (hepatitis B surface antigen positive with HBV DNA >1×10³ copies/mL; HCV RNA >1×10³ copies/mL);
* Human immunodeficiency virus (HIV) infection (HIV antibody positive);
* History or concurrent presence of other malignancies (except for effectively controlled non-melanoma skin basal cell carcinoma, in situ carcinoma of the breast/cervix, and other malignancies effectively controlled without treatment in the past five years);
* Presence of primary or secondary central nervous system (CNS) lymphoma or a history of CNS lymphoma at enrollment;
* Pregnant or lactating women, and patients of childbearing potential unwilling to use contraception;
* Requirement for systemic corticosteroid therapy or other immunosuppressive therapy due to a medical condition within 14 days before the start of study treatment [topical use (ocular, intra-articular, intranasal, and inhaled corticosteroids with minimal systemic absorption) is permitted; short-term (≤7 days) corticosteroid use for prophylaxis (e.g., contrast agent allergy) or treatment of non-autoimmune conditions (e.g., delayed hypersensitivity due to contact allergens) is permitted];
* Other conditions deemed by the investigator to be unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-02-25 (Estimated); Primary Completion 2027-10-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Complete response rate (CRR) | every 2 cycles, up to 4 cycles (each cycle is 21 days)
  Response is assessed according to the lugano criteria.

SECONDARY OUTCOMES:
Objective response rate (ORR) | every 2 cycles, up to 4 cycles (each cycle is 21 days)
  Response is assessed according to the lugano criteria.
Duration of response (DoR) | 2 years
  The time from the first assessment of CR or PR for the tumor to the first assessment of recurrence or PD or death from any cause.
Progression-free survival (PFS) | 2 years
  PFS was defined as the time between randomization and the first date of progression, relapse, or death from any cause.
Overall survival (OS) | 2 years
  From the date of randomization to date of death, irrespective of cause.
Adverse events (AEs) | From the start of treatment to 28 days after the end of treatment.
  The incidence, type, and severity of adverse events (graded according to CTCAE v5.0), and their relationship to the study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xu, Principal Investigator — The first Affiliated Hospital of Nanjing Medical University(JiangSu Province Hospital); Jinhua Liang, Principal Investigator — The first Affiliated Hospital of Nanjing Medical University(JiangSu Province Hospital)

IPD SHARING:
Plan to Share IPD: No